CLINICAL TRIAL: NCT01252511
Title: Surgical Treatment of Severe Obesity by Roux-en-Y Gastric Bypass: a Randomized Prospective Study on the Effect of Reciprocal Changes in Y-limb Lengths on Intestinal Absorption of Dietary Fat, Protein and Carbohydrate.
Brief Title: Determinants of Fat Malabsorption After Roux-en-Y Gastric Bypass
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 010-271
Record Dates: First submitted 2010-12-01; First posted 2010-12-03 (Estimated); Last update posted 2019-05-17 (Actual); Status verified 2016-01

CONDITIONS: Severe Obesity
Keywords: Malabsorption after RYGB; Fat Malabsorption and maldigestion; Obesity surgery; Bariatric surgery
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- long biliopancreatic limb, 75 cm (Active Comparator)
  Interventions: Procedure: RYGB for surgical treatment of severe obesity
- long Roux limb, 150 cm (Active Comparator)
  Interventions: Procedure: RYGB for surgical treatment of severe obesity

INTERVENTIONS:
Procedure: RYGB for surgical treatment of severe obesity — Twenty severely obese patients who have been scheduled to receive long limb RYGB will be enrolled in the study. By randomization, 10 patients will have a biliopancreatic limb that includes 40 cm of jejunum and a Roux limb that contains 150 cm of jejunum. The other 10 patients will receive a biliopancreatic limb that contains 75 cm of jejunum and a Roux limb of 115 cm.

SUMMARY:
The purpose of this study is to determine whether or not the length of the biliopancreatic limb of the Roux-en-Y anastamosis plays a critical role in the development of malabsorption after gastric bypass for treatment of severe obesity.

DETAILED DESCRIPTION:
Successful surgical treatment of severe obesity by RYGB is believed to require a procedure that (a) restricts the consumption of combustible food energy, and (b) reduces the intestinal absorption of food energy that is consumed. However, with RYGB operations that are currently employed, many patients do not develop the malabsorption they presumably require to produce good long term control of their body weight. It is important to find a way to do RYGB surgery in a way that consistently produces a moderate degree of fat malabsorption.

Patients who are scheduled to receive a RYGB for treatment of severe obesity will be randomly assigned to receive 2 variations of the standard operation. The stomach and duodenal bypass, and the creation of a small gastric pouch will be exactly the same for all patients. There will be differences in the two jejunal limbs which create the Roux-en-Y anastomosis. In Procedure A, the Roux limb length will be 150 cm, and the biliopancreatic limb will contain 40 cm of jejunum. In Procedure B, the Roux limb length will be 110 cm and the biliopancreatic limb will contain 80 cm of jejunum. The total length of jejunum in both limbs is 190 cm in both procedures. Thus, the only difference between procedures A and B is that B procedure has a larger percentage of jejunum in the biliopancreatic limb (80/190=42%) than procedure A (40/190 = 21%). A total of 20 patients will be studied, 10 with each procedure. Before and after RYGB, the patients will be studied in a clinical research laboratory. Dietary intake and intestinal absorption of fat, protein, carbohydrate and combustible energy will be measured by metabolic balance techniques for 72 hours. We hypothesize that fat malabsorption after bypass will be greater and more consistent in patients who receive the longer biliopancreatic limb than in the patients who receive the longer Roux limb.

ELIGIBILITY:
Inclusion Criteria:

* Patients with severe obesity (BMI equal to or greater than 50) who have been scheduled to receive Roux-en-Y gastric bypass.

Exclusion Criteria:

* Previous abdominal surgery, chronic diarrhea, and severe constipation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-01; Primary Completion 2014-08 (Actual); Study Completion 2017-01-14 (Actual)

PRIMARY OUTCOMES:
Selective fat malabsorption | 1 year after RYGB surgery
  To learn how to create an operation resulting in the predominance of fat malabsorption over protein malabsorption.

CONTACTS AND LOCATIONS:
Overall Officials: John S Fordtran, MD, Principal Investigator — Baylor Health Care System
Locations (1):
- Baylor University Medical Center, Dallas, Texas, United States